CLINICAL TRIAL: NCT04424056
Title: An Open Randomized Therapeutic Trial Using ANAKINRA, TOCILIZUMAB Alone or in Association With RUXOLITINIB in Severe Stage 2b and 3 of COVID19-associated Disease
Brief Title: A Trial Using ANAKINRA, TOCILIZUMAB Alone or in Association With RUXOLITINIB in Severe Stage 2b and 3 of COVID19-associated Disease
Acronym: INFLAMMACOV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-23
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Interleukin 1 Receptor Antagonist Protein; ruxolitinib; tocilizumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anakinra +/- Ruxolitinib (Experimental): Anakinra +/- Ruxolitinib
  According to clinical stage (gradual strategy):
  Stage 2b or 3 : Anakinra +/- ruxolitinib depending of evolution; Advanced stage 3 : Anakinra and Ruxolitinib
  Interventions: Drug: Anakinra +/- Ruxolitinib (stages 2b/3); Drug: Anakinra and Ruxolitinib (Advanced stage 3)
- Tocilizumab +/- Ruxolitinib (Experimental): Tocilizumab +/- Ruxolitinib
  According to clinical stage (gradual strategy):
  Stage 2b or 3 : Tocilizumab +/- ruxolitinib depending of evolution; Advanced stage 3: Tocilizumab +ruxolitinib
  Interventions: Drug: Tocilizumab +/- ruxolitinib (stages 2b/3); Drug: Tocilizumab and Ruxolitinib (Advanced stage 3)
- Standard of care (Active Comparator): Treatment with drugs or procedures in routine clinical practice
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Anakinra +/- Ruxolitinib (stages 2b/3) — administration of Anakinra +/- ruxolitinib, depending of evolution
  Arms: Anakinra +/- Ruxolitinib
Drug: Anakinra and Ruxolitinib (Advanced stage 3) — administration of Anakinra and ruxolitinib
  Arms: Anakinra +/- Ruxolitinib
Drug: Tocilizumab +/- ruxolitinib (stages 2b/3) — administration of Tocilizumab +/- ruxolitinib, depending of evolution
  Arms: Tocilizumab +/- Ruxolitinib
Drug: Tocilizumab and Ruxolitinib (Advanced stage 3) — administration of Tocilizumab and Ruxolitinib
  Arms: Tocilizumab +/- Ruxolitinib
Other: Standard of care — Treatment with drugs or procedures in routine clinical practice
  Arms: Standard of care

SUMMARY:
COVID19-associated disease may have different clinical aspects classified in 3 stages. Some patients initially presenting with a non-hypoxemic viral pneumonia (stage 2a) may evolve toward a more severe stage 2b or 3 (acute respiratory distress syndrome, ARDS) around the 7th or 10th day of evolution, with a severe biological inflammatory syndrome (CRP>200 mg/l), and some times more severe complications such as acute renal insufficiency, consumptive coagulopathy or shock, requiring increasing oxygen therapy, ICU admission, invasive mechanical ventilation and possibly leading to death. This detrimental evolution is due to a host-derived "cytokine storm" with a great excess of circulating inflammatory cytokines. In animal models of ARDS complicating coronavirus or influenza virus infection, the cytokine storm has been linked to hyperactivation of the NLRP3 inflammasome. NLRP3 constitutes an intracellular protein platform which is responsible for caspase1 activation and processing of interleukin (IL)-1beta and IL-18 . IL-1b is a major proinflammatory cytokine which induces IL-6, whereas IL-18 is an inducer of interferon gamma (IFNg) production by Th-1 lymphocytes. A blood IL-1/IL-6 signature can be defined by increased neutrophilia and CRP concentrations, whereas an IL-18/IFNg signature is characterized by severe hyperferritinemia, consumptive coagulopathy and cytopenia. A majority of patients with COVID-19 infections seems to have an IL-1/IL-6 signature, evolving in the more severe forms toward an IL-18/IFNg signature, mimicking cytokine profiles observed in other inflammatory diseases such as Still's disease or hemophagocytic syndromes. In Still's disease, therapeutic inhibition of IL-1 or IL-6 has proven to be very efficient strategies. During hemophagocytic syndromes, inhibition of IFNg is effective in humans notably through blockade of its receptor signalization, using the JAK kinase inhibitor ruxolitinib.

Following this strategy, we propose to use biological drugs currently available for inhibition of IL-1 (anakinra), IL-6 (tocilizumab) or IFNg signaling (ruxolitinib) in the severe forms of COVID19-associated disease. Our hypothesis is that IL-1, IL-6 or JAK kinase inhibition will allow:

1. to prevent stage 2b worsening and the need to be admitted in ICU, by decreasing oxygen-requirement and systemic inflammation
2. to improve stage 3 and extremely severe stage 3, allowing invasive mechanical ventilation weaning, improving multi-system organ dysfunction, leading to a faster ICU exit.

We propose an open randomized therapeutic trial (1/1/1) on 216 patients with severe stage 2b and 3 of the disease

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 year up to 75 year-old maximum
* Eligible for resuscitation care in UCI
* with proven infection with COVID-19, using at least one positive pharyngeal polymerase chain reaction (PCR) test
* COVID19 infection pneumonia at

  * Stage 2b: Hypoxemic pneumonia (respiratory rate >30/min, Sat O2<90 mm Hg in ambient air) associated with a marked biological inflammatory syndrome (CRP>150mg/l) - or Stage 3: ARDS defined by a mechanically ventilated patient with a PaO2/FiO2 ratio < 300 for more than 24 hours.
  * or Advanced Stage 3: moderate to severe ARDS (PaO2/FiO2 < 200 to PEEP of at least 8 cmH2O) on invasive mechanical ventilation associated with another organ failure or syndrome among : 1) Shock with norepinephrine dosage > 3 mg/hour, 2) Acute renal oligo-anuric failure or requiring extra-renal lavage, 3) Hepatocellular failure or coagulopathy with factor V < 50%, 4) Myocarditis causing acute heart failure and/or shock. , 5) Hemophagocytic syndrome, 6) Hyperferritinemia > 5000 ng/mL

Exclusion Criteria:

* Patients younger than 18 or older than 75 year-old,
* Pregnant or breastfeeding woman
* Patient for whom measures of therapeutic limitations have been issued (non-admission to intensive care unit)
* Patients treated with immunosuppressant/immunomodulators (Not only the concomitant administration of the following drugs prohibited in the protocol: other JAK inhibitors, corticosteroids, IL6 inhibitors).
* Patient already included in another interventional therapeutic trial
* Use of chronic oral corticosteroids > 10 mg prednisone equivalent per day for non-COVID-19 related disease
* Uncontrolled autoimmune disease
* Patients with active, suspected or known active systemic bacterial, viral (excluding COVID-19) or fungal infections that are not controlled (not only HIV, HBV or HCV infection and untreated bacterial or mycotic infection)
* Patients with severe pre-existing uncontrolled organ dysfunction (heart, liver or kidney failure) not related to COVID-19

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation free days at D28 | 28 days
  number of days living without mechanical ventilation at D28

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No